CLINICAL TRIAL: NCT00420264
Title: Feasibility of Using Gynecare Thermachoice III in the Office Setting Without Conscious Sedation
Brief Title: ThermaChoice III Under Local Sedation in the Office Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Female Pelvic Medicine & Urogynecology Institute of Michigan (Other)
Collaborators: Ethicon, Inc. (Industry)
Responsible Party: Jason B. Bennett, MD, Female Pelvic Medicine & Urogynecology Institute of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: ThermaChoice III
Record Dates: First submitted 2007-01-10; First posted 2007-01-11 (Estimated); Last update posted 2013-08-14 (Estimated); Status verified 2013-08

CONDITIONS: Heavy Uterine Bleeding

INTERVENTIONS:
Device: Uterine Ablation — Uterine Ablation in the office setting to see if the procedure is tolerated w/o sedation

SUMMARY:
Investigational study to determine if an endometrial ablation for heavy uterine bleeding, can be tolerated in the office setting without the use of intravenous medication.

DETAILED DESCRIPTION:
A safe and effective treatment , called endometrial ablation, has been used in a hospital setting under general anesthesia for the treatment of heavy uterine bleeding. This study will evaluate if patients would tolerate the same procedure in an office setting using local anesthetics and common pain medication. This study will include twenty patients.

ELIGIBILITY:
Inclusion Criteria:

* Heavy uterine bleeding

Exclusion Criteria:

* Uterine or cervical cancer
* Unable to tolerate office hysteroscopy
* Uterine fibroid tumors that distort endometrial cavity
* Uterine cavity greater than 12 cm
* Patients with hyperplasia or premalignant changes of the endometrium
* Active genital or urinary tract infections
* Intrauterine device
* Pregnant or want to become pregnant

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2005-11; Primary Completion 2008-06 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Tolerability of Uterine Ablation in the office setting | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Jason B Bennett, MD, Principal Investigator — Grand Valley Gynecologists, PC
Locations (1):
- Grand Valley Gynecologists, PC, Grand Rapids, Michigan, United States